CLINICAL TRIAL: NCT01600118
Title: Effect of Low-energy Extracorporeal Shock Waves on Periodontal and Endodontic Parameters
Brief Title: Effect of Shock Waves on Dental Parameters
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Frank Falkensammer, DMD,DMS, DMD,DMS, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESWT1
Record Dates: First submitted 2012-05-14; First posted 2012-05-16 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Tooth Stability; Blood Flow
Keywords: tooth mobility; periodontal status; irregularity index; pulpal blood flow
MeSH Terms: conditions — Tooth Mobility | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ESWT (Active Comparator): Extracorporeal shockwave therapy
  Interventions: Device: Extracorporeal shockwave therapy
- ESWT Placebo (Placebo Comparator): No extracorporeal shockwave therapy
  Interventions: Device: No extracorporeal shockwave

INTERVENTIONS:
Device: Extracorporeal shockwave therapy — 1000 impulses
  Other Names: Orthogold 100 MTS
  Arms: ESWT
Device: No extracorporeal shockwave — 0 impulses, acoustic effect
  Arms: ESWT Placebo

SUMMARY:
This randomized clinical trial investigates the effect of the extracorporeal shockwave therapy (ESWT) on periodontal and endodontical parameters. The ESWT is a scientifically approved non invasive method to influence bone turnover and tissue regeneration. The hypotheses of this trial are that ESWT increases the periodontal stability of orthodontically aligned teeth as well as increase the blood flow. Increasing the periodontal stability would reduce the retention phase, relapse risk and accelerate the rehabilitation of the surrounding tissues.

ELIGIBILITY:
Inclusion Criteria:

* healthy patients which don´t fulfill the exclusion criteria

Exclusion Criteria:

* diseases (syndroms, infections,...) which influence the bone turnover and blood flow
* medication, which influences the bone turnover and blood flow
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-09; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
periodontal stability of orthodontically aligned teeth | 6 months

SECONDARY OUTCOMES:
pulpal blood flow | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Bernhard Gottlieb University clinic of Dentistry, Vienna, Vienna, Austria

REFERENCES:
- [Result] Sathishkumar S, Meka A, Dawson D, House N, Schaden W, Novak MJ, Ebersole JL, Kesavalu L. Extracorporeal shock wave therapy induces alveolar bone regeneration. J Dent Res. 2008 Jul;87(7):687-91. doi: 10.1177/154405910808700703. PMID 18573992
- [Result] Martini L, Giavaresi G, Fini M, Torricelli P, de Pretto M, Schaden W, Giardino R. Effect of extracorporeal shock wave therapy on osteoblastlike cells. Clin Orthop Relat Res. 2003 Aug;(413):269-80. doi: 10.1097/01.blo.0000073344.50837.cd. PMID 12897619